CLINICAL TRIAL: NCT03940599
Title: Investigating the Impact of Self-monitoring Feedback for Health Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2000021910
Record Dates: First submitted 2019-04-29; First posted 2019-05-07 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fitbit with visible screen (Experimental): The first group will receive a FitBit with the screen visible, displaying their daily step count (the Step-Counter group).
  Interventions: Device: step counter
- Scale group (Experimental): The second will receive a BodyTrace scale that will display and record their weight in kilograms and a FitBit with the screen covered as it was for the run-in period so their physical activity can be measured, but the only feedback they will receive is from the scale (the Scale group).
  Interventions: Device: weight scale; Device: step counter with screen covered
- Step counter and scale (Experimental): The third group will receive a BodyTrace scale and a FitBit with the screen visible (the Step-Counter and Scale group).
  Interventions: Device: step counter; Device: weight scale
- Fitbit with screen covered (Sham Comparator): The remaining 5 participants will serve as normal controls and continue wearing the FitBit with the screen covered as it was during the run in period for the duration of follow up.
  Interventions: Device: step counter with screen covered

INTERVENTIONS:
Device: step counter — Fitbit
  Arms: Fitbit with visible screen; Step counter and scale
Device: weight scale — BodyTrace weight scale
  Arms: Scale group; Step counter and scale
Device: step counter with screen covered — Fitbit with screen covered
  Arms: Fitbit with screen covered; Scale group

SUMMARY:
Investigating the impact of self-monitoring feedback for health behaviors

DETAILED DESCRIPTION:
Obesity is highly prevalent in Samoa, where a 2010 study estimated that 64.6% of adult females were obese, according to Polynesian BMI cut offs (BMI ≥32.0 kg/m2).1,2 Interventions designed to increase physical activity or facilitate weight loss often include a self-monitoring component, but these intervention programs have not yet been tested in the Samoan setting. The goal of this project is to pilot test such an approach.

The specific aims of this study are:

1. To investigate the acceptability and feasibility of self-monitoring of physical activity and weight through the introduction of step counting devices (FitBit Zips) and scales (BodyTrace).
2. To measure any changes that occur in participants' health, health behaviors related to diet and physical activity, or conceptions of health (including self-efficacy and perceptions of weight) over the study period.

ELIGIBILITY:
Inclusion Criteria:

* Samoan ethnicity (measured by their having four Samoan grandparents)
* 31.5 - 40 years of age
* Physically inactive - defined using the World Health Organization (WHO) definition of inactivity and the WHO Global Physical Activity Questionnaire
* Motivated and ready to make behavior changes - defined using the Physical Activity Stages of Change framework (contemplation or preparation phase)18
* Not pregnant or planning to become pregnant during the 5-week study period - self-reported at baseline
* Weigh less than 180 kg - based on measured weight at baseline. This restriction is due to the maximum weight of the BodyTrace scales used in the intervention.
* No medical condition preventing physical activity or making participation inadvisable. These conditions will be measured based on self-report of doctor diagnoses and include: hypertension, heart attack, heart disease, stroke, uncontrolled Type 2 diabetes, non-skin cancer diagnosis, dialysis, or a diagnosed eating disorder. Participants will also be excluded if they have had significant (>10 kg) self-reported weight loss in the last 6 months.

Exclusion Criteria:

* If participant does not fit the requirements above

Ages: 31 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The target population for this study are healthy, Samoan women between the ages of 31.5 and 40
Enrollment: 44 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Baseline Weight measure | baseline
  This visit will take place on the same day as recruitment, after participants have completed the Village-Based Screening. Eligible participants will be flagged based on their responses to the screening questionnaire, at which point they will be informed of this additional project, complete an eligibility questionnaire, and, if interested in participating, give informed consent. At this baseline visit, they will receive a FitBit Zip with the screen covered so that they are not able to see any of the recorded information. The screen will be sealed such that the researcher will know if the participant has broken through to check the screen. Contact information will also be collected and a visit scheduled for one week later.
Weight measure - randomization | 1 week
  The participant will then complete a one week run in period to establish their baseline physical activity as measured by the FitBit. Participants will not be informed of their measured physical activity for this week and the screen will remain covered so that they are not receiving feedback from the device. After this period, the first home visit will take place. All participants will complete additional questionnaires at this time that will include information about their current health behaviors, their conceptions of their health (including their self-reported health status, self efficacy, health locus of control, and body image), and an estimate of their weight and perceived weight category (underweight, normal, overweight, or obese).
Psychological Indicators of Health questionnaire | 1 week
  All participants will complete additional questionnaires at this time that will include information about their current health behaviors, their conceptions of their health (including their self-reported health status, self efficacy, health locus of control, and body image), and an estimate of their weight and perceived weight category (underweight, normal, overweight, or obese).
Weight measure synching | 2 weeks
  The next visit will occur two weeks later, at the midpoint of the four week follow up period with the self-monitoring devices. This visit will not involve any further questionnaires and will occur for the purpose of syncing physical activity data from the FitBit, which only stores physical activity data for 23 total days.
Weight measure final | 5 weeks
  The final visit will occur two weeks later, after the full four weeks of follow up with the devices. This visit occurs at week 5 of the study, including the one week run in period. At this point participants will repeat all of the questionnaires that they previously completed, as well as having their height and weight measured again. They will also complete added questions related to changes in their health behaviors over the past month of the follow up period. All participants will also complete a semi structured, qualitative interview to capture their experience of using the self-monitoring devices. These interviews are optional. The interview will include questions about what they did or did not like about the devices, how they felt about the feedback they were receiving, and how it may have influenced their thinking and behaviors. In addition, they will keep the device.
Psychosocial Indicators of Health final questionnaire | 5 weeks
  This visit occurs at week 5 of the study, including the one week run in period. At this point participants will repeat all of the questionnaires that they previously completed, as well as having their height and weight measured again. They will also complete added questions related to changes in their health behaviors over the past month of the follow up period. All participants will also complete a semi structured, qualitative interview to capture their experience of using the self-monitoring devices. These interviews are optional. The interview will include questions about what they did or did not like about the devices, how they felt about the feedback they were receiving, and how it may have influenced their thinking and behaviors. In addition, they will keep the device.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Kocher, Principal Investigator — Yale School of Public Health
Locations (1):
- Olaga Research Laboratory - Ministry of Health, Apia, Samoa